CLINICAL TRIAL: NCT01519466
Title: Impact of a built-in Insulin Calculator Feature on Diabetes Control - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADC-PMR-INX-11012
Record Dates: First submitted 2012-01-06; First posted 2012-01-27 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; SMBG; Insulin calculator
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): Subjects will use a FreeStyle InsuLinx blood glucose meter during the study
  Interventions: Device: FreeStyle InsuLinx
- Control (Other): Subjects will use a FreeStyle Freedom Lite blood glucose meter during the study.
  Interventions: Device: FreeStyle Freedom Lite

INTERVENTIONS:
Device: FreeStyle InsuLinx — FreeStyle InsuLinx is a blood glucose meter with a built-in insulin calculator feature.
  Arms: Intervention
Device: FreeStyle Freedom Lite — FreeStyle Freedom Lite is a blood glucose meter
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the effect of using FreeStyle InsuLinx (a blood glucose meter with a built-in insulin calculator) on glucose control in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes on MDI (3 or more insulin injections per day (U100 insulin)) for at least 1 year and insulin adjusting
* HbA1c between 7.0% and 9.5% (53 to 80 mmol/mol) inclusive
* Age 18 and over
* In the investigator's opinion, thought technically capable of using masked CGM
* Subject self reporting a minimum of 21 SMBG tests per week prior to study enrolment
* Willing to perform a minimum of 4 SMBG tests per day during study

Exclusion Criteria:

* Subject has any concomitant disease or condition that, in the investigator's opinion, may compromise patient safety
* Subject is participating in another study of a glucose monitoring device / drug that could affect glucose measurements / management
* Subject is pregnant / planning to become pregnant within the planned study timeline
* Subject is known to require a dose of more than 50 units of U100 insulin in any one bolus injection
* Subject is currently on an insulin pump
* Subject is currently using the FreeStyle InsuLinx
* Subject is currently using the FreeStyle Freedom Lite
* Subject is currently using CGM
* Subject has an allergy to medical grade adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Michaela Diamant, Principal Investigator — VU University Medical Centre (VUMC)
Locations (4):
- Germany (3):
  - Diabetes Zentrum Mergentheim, Bad Mergentheim
  - Diabetes-Zentrum für Kinder und Jugendliche, Hanover
  - Institut für Diabetes - Technology Forschungs - und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm
- VU University Medical Centre (VUMC), Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 55 subjects consented and enrolled into the study. Six of these withdrew before randomisation or failed screening. Forty-nine (49) subjects were randomised and completed the study.
Groups:
- FreeStyle InsuLinx: Subjects will use a FreeStyle InsuLinx blood glucose meter during the study
  FreeStyle InsuLinx: FreeStyle InsuLinx is a blood glucose meter with a built-in insulin calculator feature.
- FreeStyle Freedom Lite: Subjects will use a FreeStyle Freedom Lite blood glucose meter during the study.
  FreeStyle Freedom Lite: FreeStyle Freedom Lite is a blood glucose meter
Period: Overall Study
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite
Started | 33 | 16
Completed | 33 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 55 subjects consented and enrolled into the study. Six of these withdrew before randomisation or failed screening. Forty-nine (49) subjects were randomised and completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (15.2) | 43.4 (16.7) | 44.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 17 | 9 | 26
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 4 | 12
  Germany | 25 | 12 | 37
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 26.6 (3.6) | 26.4 (4.4) | 26.5 (3.8)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 18.8 (14.1) | 14.6 (8.0) | 17.4 (12.5)
Screening HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 61.7 (7.7) | 64.8 (6.8) | 62.7 (7.5)
Screening HbA1c [Mean (Standard Deviation); unit: Percentage of Glycosylated Haemoglobin] | 7.8 (0.7) | 8.1 (0.6) | 7.9 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Time in Target Blood Glucose Range
Description: Masked continuous glucose monitoring data will be collected for two weeks at the start of the study and 2 weeks at the end of the study. Analysis will assess the difference between the assessment and baseline phase for the intervention group. Target blood glucose range is 3.9 to 10.0mmol/l (70 to 180mg/dL)
Time Frame: Day 1-15 compared with Day 60-74
Population: One FreeStyle InsuLinx group subject was excluded from the analysis due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite
Number analyzed (Participants) | 32 | 16
hours per day
  Baseline | 15.28 (2.76) | 15.31 (3.15)
  Final | 14.56 (2.99) | 14.14 (2.36)
Statistical Analysis 1: Comparison: FreeStyle InsuLinx; Test type: Superiority or Other; p = 0.0926, t-test, 2 sided; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.55 to 0.12], Standard Deviation 2.32
Statistical Analysis 2: Comparison: FreeStyle Freedom Lite; Test type: Superiority or Other; Mean Difference (Final Values) = -1.17, Standard Deviation 2.97

2. Secondary Outcome: HbA1c
Description: HbA1c will be tested at baseline (day 1) and then again at end of study (approximately day 74).
  The percentage of glycosylated hemoglobin in Diabetes Control and Complications Trial (DCCT) units was standardized to the newer International Federation of Clinical Chemistry (IFCC) units (mmol/mol).
Time Frame: Day 1 compared with Day 74
Population: One FreeStyle InsuLinx group subject was excluded from the analysis due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: Percentage of Glycosylated Haemoglobin
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite
Number analyzed (Participants) | 32 | 16
Percentage of Glycosylated Haemoglobin
  Baseline | 7.87 (0.76) | 8.07 (0.76)
  Final | 7.78 (0.58) | 7.98 (0.69)
Statistical Analysis 1: Comparison: FreeStyle InsuLinx; Test type: Superiority or Other; p = 0.3251, t-test, 2 sided; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.27 to 0.09], Standard Deviation 0.49
Statistical Analysis 2: Comparison: FreeStyle Freedom Lite; Test type: Superiority or Other; Mean Difference (Final Values) = -0.09, Standard Deviation 0.51

3. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQc) Scores From Day 1 to Day 60.
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale (-3 to +3). The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied).
  There is one question to assess the change in satisfaction with perceived frequency of Hypoglycaemia and one question to assess change satisfaction with perceived frequency of Hyperglycaemia. Each question is rated on a 7-point Likert scale (-3 to +3), -3 (much less satisfied) to +3 (much more satisfied).
  The 95% confidence intervals for the FreeStyle InsuLinx group DTSQc scores was calculated using a one-sample t-test.
Time Frame: Day 60 compared to day 1
Population: One FreeStyle InsuLinx group subject was excluded from the analysis due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite
Number analyzed (Participants) | 32 | 16
Units on a scale
  Hyperglycaemia | 0.13 (1.26) | -0.25 (1.53)
  Hypoglycaemia | -0.31 (1.03) | 0.13 (1.02)
  Treatment Satisfaction | 4.36 (6.53) | 2.94 (7.92)
Statistical Analysis 1: Comparison: FreeStyle InsuLinx; Hyperglycaemia, glucose above 10mmol/l (180mg/dL); Test type: Superiority or Other; p = 0.5798, t-test, 2 sided; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.33 to 0.58], Standard Deviation 1.26
Statistical Analysis 2: Comparison: FreeStyle InsuLinx; Hypoglycaemia, glucose below 3.9mmol/l (70mg/dL); Test type: Superiority or Other; p = 0.0960, t-test, 2 sided; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.68 to 0.06], Standard Deviation 1.03
Statistical Analysis 3: Comparison: FreeStyle InsuLinx; Treatment Satisfaction; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided; Mean Difference (Final Values) = 4.36, 95% CI 2-sided [2.01 to 6.71], Standard Deviation 6.53

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrolment to completion by last subject (up to 3 months).
Arm/Group | FreeStyle InsuLinx | FreeStyle Freedom Lite
Serious Adverse Events (participants affected / at risk) | 3/33 | 2/16
Other Adverse Events (participants affected / at risk) | 8/33 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FreeStyle InsuLinx (N=33) | FreeStyle Freedom Lite (N=16)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gingiva abcess (Infections and infestations) | 0 (0) | 1 (1)
Fractured Metacarpus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sensor tip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FreeStyle InsuLinx (N=33) | FreeStyle Freedom Lite (N=16)
Cold (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Endocrine disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days